CLINICAL TRIAL: NCT02782624
Title: Relative Bioavailability of 5 mg BI 10773 Administered Twice Daily Compared to 10 mg BI 10773 Given Once Daily After Multiple Oral Doses in Healthy Male and Female Volunteers (an Open-label, Randomised, Crossover, Clinical Phase I Study)
Brief Title: Relative Bioavailability of BI 10773 Administered Twice Daily Compared BI 10773 Given Once Daily After Multiple Oral Doses in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1276.9; 2009-012524-90 (EudraCT Number: EudraCT)
Record Dates: First submitted 2016-05-23; First posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin

ARMS (2):
- Treatment A: Empagliflozin (Experimental): 5 mg bid
  Interventions: Drug: Empagliflozin
- Treatment B: Empagliflozin (Experimental): 10 mg qd
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — 5 days of treatment with 5 mg BI 10773 bid until steady state
  Arms: Treatment A: Empagliflozin
Drug: Empagliflozin — 5 days of treatment with 10 mg BI 10773 qd until steady state
  Arms: Treatment B: Empagliflozin

SUMMARY:
To investigate the influence of different dosage regimen (5 mg twice daily versus 10 mg once daily) on the steady state pharmacokinetics and pharmacodynamics of BI 10773 administered orally

ELIGIBILITY:
Inclusion criteria:

- Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests

* Age = 18 and Age = 50 years
* BMI = 18.5 and = 29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders 6. History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs within one month or less than 10 half-lives of the respective drug prior to first study drug administration except if a relevant interaction can be ruled out
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (average consumption of more than 20 g/day in females and 30 g/day in males)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to the start of study)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

For female subjects:

* Positive pregnancy test, pregnancy or planning to become pregnant during the study or within 1 month after study completion
* No adequate contraception during the study and until 1 month after study completion, i.e. not any of the following: implants, injectables, combined oral contraceptives, IUD A record of all subjects screened, in- or excluded, will be maintained. (intrauterine device), sexual abstinence for at least 1 month prior to enrolment, vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (including hysterectomy). Females, who do not have a vasectomised partner, are not sexually abstinent or surgically sterile will be asked to use an additional barrier method (e.g. condom, diaphragm with spermicide)
* Lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
AUC (area under the concentration-time curve of the analyte in plasma) - AUCt,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval t) for 10 mg BI 10773 QD. | up to 168 hours
AUC (area under the concentration-time curve of the analyte in plasma) - AUC0-24,ss (area under the concentration-time curves of the analyte in plasma at steady-state over two dosing intervals) for 5 mg BI 10773 BID after the morning dose on Day 5. | up to 168 hours
AUCt,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval t) of BI 10773. | up to 168 hours
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval t) of BI 10773. | up to 168 hours

SECONDARY OUTCOMES:
C12,N (concentration of analyte in plasma at 12 hours post-drug administration after administration of the Nth dose for the BID regimen) of BI 10773. | up to 168 hours
C24,N (concentration of analyte in plasma at 24 hours post-drug administration after administration of the Nth dose for the QD regimen) of BI 10773. | up to 168 hours
Cmin,ss (minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval t) of BI 10773 | up to 168 hours
Cavg (average concentration of the analyte in plasma at steady state) of BI 10773 | up to 168 hours
¿z,ss (terminal half-life of the analyte in plasma at steady state) of BI 10773 | up to 168 hours
t½,ss (terminal half-life of the analyte in plasma at steady state) of BI 10773 | up to 168 hours
tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state over a uniform dosing interval t) of BI 10773. | up to 168 hours
MRTpo,ss (mean residence time of the analyte in the body at steady state after oral administration) of BI 10773. | up to 168 hours
CL/F,ss (apparent clearance of the analyte in the plasma after extravascular administration at steady state) of BI 10773. | up to 168 hours
Vz/F,ss (apparent volume of distribution during the terminal phase tau z at steady state following extravascular administration) of BI 10773. | up to 168 hours
PTF (percentage peak-trough fluctuation) | up to 168 hours

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1276.9.1 Boehringer Ingelheim Investigational Site, Biberach, Germany